CLINICAL TRIAL: NCT05398159
Title: Safety and Efficacy of Trim II for Non-invasive Lipolysis and Circumference Reduction of Abdomen
Brief Title: Trim II for Noninvasive Lipolysis and Circumference Reduction of Abdomen.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DO609924A
Record Dates: First submitted 2022-05-17; First posted 2022-05-31 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Circumference Reduction of Abdomen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- treatment (Experimental): 3 bi-weekly treatments
  Interventions: Device: Trim II

INTERVENTIONS:
Device: Trim II — Eligible subjects will receive 3 bi-weekly treatments (once in 2 weeks) with Trim II hands-free applicator belt according to the study protocol.
  Trim II hands-free applicator composed of 4 units applied to the abdominal area, using a single-use belt.
  Each treatment duration will be 45-60 minutes. Study duration for each subject is approximately 6 months (including screening, 3 treatments and 2 follow-up visits at 1 and 3 months post last treatment).

SUMMARY:
At least 90 female and male subjects, from 6 investigational sites, aged 18-70 seeking non-invasive lipolysis and circumference reduction of abdomen will be enrolled. Eligible subjects will receive 3 bi-weekly treatments (once in 2 weeks) with Trim II hands-free applicator belt according to the study protocol.Study duration for each subject is approximately 6 months (including screening, 3 treatments and 2 follow-up visits at 1 and 3 months post last treatment).

DETAILED DESCRIPTION:
The goal of this prospective study is to evaluate Safety and Efficacy of Trim II for Non-invasive Lipolysis and Circumference Reduction of Abdomen.

The main questions are :

* Efficacy of the Trim II treatment for lipolysis and abdominal circumference reduction.
* Safety of the Trim II treatment for lipolysis and abdominal circumference reduction

Eligible subjects will receive 3 bi-weekly treatments (once in 2 weeks) with Trim II hands-free applicator belt according to the study protocol.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects, aged 18-70.
* BMI≤ 30.
* Subjects seeking non-invasive lipolysis and circumference reduction of abdomen
* Female should not be pregnant or lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrolment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
* In addition, negative urine pregnancy test as tested before each treatment and at the last visit for women with childbearing potential (e.g. not menopause).
* General good health confirmed by medical history and skin examination of the treated area.
* The subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side effects, and sign the Informed Consent Form, including permission to use photography.
* The subjects should be willing to comply with the study procedure and schedule, including the follow up visits, and will refrain from using any other abdominal treatment methods during the entire study period.

Exclusion Criteria:

* - Active electrical implant/device in any region of the body, including pacemaker or internal defibrillator
* Permanent implant in the treated area such as metal plates, screws or silicon, metal piercing or other.
* Current or history of skin cancer, or current condition of any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders, sensory disturbances, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants except for low-dose aspirin.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV or use of immunosuppressive medications.
* Pregnancy and nursing.
* Poorly controlled endocrine disorders, such as Diabetes, or thyroid dysfunction and hormonal virilization.
* Isotretinoin (Accutane) within last 6 months.
* Any active condition in the treatment area, such as sores, Psoriasis, eczema, and rash, open lacerations, abrasions or lesions, infection in the area to be treated.
* Any surgical procedure in the treatment area within the last 12 months or before complete healing.
* Having received treatment with light, laser, RF, or other devices in the treated area within 2-3 weeks for non-ablative procedures, and 6-12 weeks for ablative fractional laser resurfacing (according to treatment severity) prior to treatment, except special recommendations.
* Use of non-steroidal anti-inflammatory drugs (NSAIDS, e.g., ibuprofen-containing agents) one week before and after each treatment session, as per the practitioner's discretion.
* As per the investigator's discretion, refrain from treating any condition which might make it unsafe for the patient.
* Participated in another investigational drug or device study or have completed the follow-up phase for any previous study less than 30 days prior to the first evaluation in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-10-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - H/K/B Cosmetic Surgery, Huntersville, North Carolina
  - Bucky Body Center, Philadelphia, Pennsylvania
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Dallas Plastic Surgery Institute, Dallas, Texas
  - Refresh Dermatology, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Labadie JG, Chilukuri S, Cohen J, Kilmer S, Lupo M, Rohrich R, Dover JS. Noninvasive Hands-free Bipolar Radiofrequency Facial Remodeling Device for the Improvement of Skin Appearance. Dermatol Surg. 2023 Jan 1;49(1):54-59. doi: 10.1097/DSS.0000000000003666. Epub 2022 Dec 8. PMID 36533797

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: 3 bi-weekly treatments
  Trim II: Eligible subjects will receive 3 bi-weekly treatments (once in 2 weeks) with Trim II hands-free applicator belts according to the study protocol.
  Each treatment duration will be 45-60 minutes.
Period: Overall Study
Arm/Group | Treatment
Started | 75
Completed | 44
Not Completed | 31

BASELINE CHARACTERISTICS:
Groups:
- Treatment: 3 bi-weekly treatments
  Trim II: Eligible subjects will receive 3 bi-weekly treatments (once in 2 weeks) with Trim II hands-free applicator belt according to the study protocol.
  Each treatment duration will be 45-60 minutes.
Arm/Group | Treatment
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: dropouts
  years | 47.6 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: dropouts
  Participants
    Female | 39
    Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 38
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants] — Population: dropouts
  participants
    United States | 44
Skin type [Count of Participants; unit: Participants] — The Fitzpatrick scale (also Fitzpatrick skin typing test; or Fitzpatrick phototyping scale) is a numerical classification schema for human skin color. Skin color classified to I, II, III, IV or V skin type. Skin type I is the lightest and V is the darkest.
  Participants
    Skin type I | 5
    Skin type II | 24
    Skin type III | 7
    Skin type IV | 5
    Skin type V | 3
    Skin type VI | 0
Body Mass Index [Mean (Standard Deviation); unit: units of kg/m2] | 24 (3.0)
Subjects Height [Mean (Standard Deviation); unit: inch] | 66.1 (4)
Subjects Weight [Mean (Standard Deviation); unit: pounds] | 149.8 (21.5)
Circumference Measurements [Mean (Standard Deviation); unit: cm] — Patients had complete baseline and 3-month follow-up data for tape measurement of circumference. There were 3 measurement points for this evaluation: widest circumference, 2 inches above umbilicus, and 2 inches below the umbilicus calculated as average.
  cm | 91.4 (7.6)
Caliper Measurements [Mean (Standard Deviation); unit: mm] — Patients had complete caliper measurements of fat thickness data for baseline and 3-month follow-up timepoints. Caliper measurements were performed on both sides of the belly button and the two measurements are assessed as averaged together
  mm | 22.9 (10.6)
Ultrasound measurements of fat thickness [Mean (Standard Deviation); unit: mm] — Two ultrasound measurements were performed at two time points (baseline and 3 months post-treatment) to measure abdominal subcutaneous fat in the area of the two measurement points.
  mm | 24.5 (5.9)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Change in Abdomen Circumference Using Tape Measurements in cm at the 3 Months Follow-up Visit Comparing to Baseline.
Description: Efficacy of the Trim II treatment for lipolysis and abdominal circumference reduction.
  Evaluation of change in abdomen circumference using tape measurements in cm at the 3 months follow-up visit comparing to baseline.
  Success criteria: Statistically significant reduction in abdominal circumference tape measurements at the 3 months follow-up visit compared to baseline
Time Frame: 3 months
Population: treatment arm
Measure: Mean (Standard Deviation); unit: CM
Arm/Group | Treatment
Number analyzed (Participants) | 44
CM | 89.5 (8.3)

2. Primary Outcome: Safety of the Trim II Treatment for Lipolysis and Abdominal Circumference Reduction.
Description: Number of participants with incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]) will be followed throughout the whole study. Observation, assessment, and recording of potential reactions by the investigator.
  Evaluations will be done immediately after each treatment and at the follow-up visits. The frequency, severity, and causality of reactions will be recorded.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Treatment
Number analyzed (Participants) | 44
participants | 2

3. Secondary Outcome: Percentage of Participants With Baseline and 3 Month Abdomen Photographs Correctly Identified by Two Blind Evaluators
Description: Success criteria: Correct identification of baseline and 3-month follow-up visit photographs of the abdomen (treatment) area in at least 70% of treated subjects by two blinded evaluators.
Time Frame: 3 months
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 44
percentage of participants | 86.4

4. Secondary Outcome: Change in Abdominal Fat Thickness Measured by Ultrasound Imaging (USI) at the 3 Months Follow-up Visit Comparing to Baseline.
Description: Success criteria: statistically significant change in fat thickness of the abdomen (treatment) area measurements at the 3 months follow-up visit compared to baseline.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Treatment
Number analyzed (Participants) | 44
mm | 21.4 (5.3)

5. Secondary Outcome: Subject's Satisfaction With Study Treatment at 3 Months Follow-up Visit.
Description: Subject's satisfaction with the therapy results was evaluated through the Subject Satisfaction Questionnaire (5-point scale). The higher the score the better the outcome. 2-Very satisfied, 1-satisfied, 0-indifferent, -1 disappointed, -2- very disappointed
Time Frame: 3 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 44
score on a scale | 0.63 [-2 to 2]

6. Secondary Outcome: Treatment Comfort During the Study Treatment.
Description: Average of comfort post treatment evaluated using the Therapy Comfort Questionnaire. Scored from-2 to +2. The higher the score the better the outcome. Average value is calculated
Time Frame: Immediately post each treatment once in 2 weeks for 6 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 44
score on a scale | 0.61 [-2 to 2]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 2/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=75)
burn (Skin and subcutaneous tissue disorders) | 1 (1)
blisters (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-03): https://cdn.clinicaltrials.gov/large-docs/59/NCT05398159/Prot_SAP_001.pdf